CLINICAL TRIAL: NCT03820999
Title: An Intervention in a Primary Healthcare Setting to Reduce Lyme Neuroborreliosis Treatment Delay
Acronym: NBdelay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Fredrikke Christie Knudtzen, Speciality Registrar, Specialist in Infectious Diseases, Principal Investigator, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCKPhDProject4
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Lyme Neuroborreliosis
Keywords: treatment delay; primary health care
MeSH Terms: conditions — Lyme Neuroborreliosis

STUDY DESIGN:
Intervention Model Description: Open label interventional study where primary Health care Physicians in areas on Funen Island, Denmark, are included if they have their practice in an area with Lyme Neuroborreliosis incidens > 4.6/100.000
Masking Description: Open label study, due to the intervention (lectures) and the criteria for receiving the intervention (Lyme neuroborreliosis incidens > 4.6/100.000), the study cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teaching arm (Experimental): The Primary Health Care physicians getting oral and written information on tick-bites and Lyme disease with focus on Lyme neuroborreliosis.
  Interventions: Other: Oral and written information on tick-bites and Lyme disease
- Passive arm (No Intervention): The Primary Health Care physicians that does not get contacted with an offer to receive oral and written information.

INTERVENTIONS:
Other: Oral and written information on tick-bites and Lyme disease — See under study arm descriptions
  Arms: Teaching arm

SUMMARY:
This study evaluates the effect of written and oral information in a primary health care setting on 1) patients referred to specialised examination for Lyme neuroborreliosis, 2) delay from patient symptom debut to treatment for Lyme neuroborreliosis, and 3) number of Borrelia serology tests from primary health care.

DETAILED DESCRIPTION:
Lyme neuroborreliosis is among the most common neuroinfections in northern Europe. Residual symptoms after treatment are a frequent problem in Lyme neuroborreliosis, and an association between the delay from symptom debut to antibiotic treatment has been established. In a previous study on Funen Island, Denmark, the delay from day of symptom debut to treatment for Lyme neuroborreliosis patients was 24 days. This considerable treatment delay did not change in the 20 years study period.

In the Danish health system, the general practitioners are the first medical professionals to see the majority of patients. They can refer patients to the hospital for further examination if indicated. Many general practitioners use Borrelia burgdorferi antibodies (igM/IgG) as a screening tool when they suspect Lyme disease or see patients with uncharacteristic symptoms. This is unfortunate, as the rash Erythema Migrans, the most common Borreliosis manifestation in Europe, is a clinical diagnosis. Only around 50% of patients have positive antibodies at time of Erythema Migrans diagnosis. Lyme neuroborreliosis is diagnosed based on symptoms and the results from the cerebrospinal fluid, and cannot be diagnosed based on serology, which only delays the time to diagnoses and treatment. The Danish guidelines on Lyme borreliosis therefore discourage general practitioners from using Borrelia serology.

In the before mentioned study from Funen Island, several patients described multiple contacts to their general practitioners, where the symptoms of Lyme neuroborreliosis were not recognized. The cardinal symptom of radicular pain was associated with a longer delay than many of the less common symptoms of Lyme neuroborreliosis.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians with a postal code in an area of Funen Island with a Lyme neuroborreliosis incidens of > 4.6/100.000
* Patients with a postal address on Funen and a positive Borrelia intrathecal antibody test (diagnostic for lyme neuroborreliosis) performed at the Department of Clinical Microbiology, Odense University Hospital from January 1st 2017 - December 31st 2020
* A Borrelia IgM/IgG serology ordered from Primary Health Care and performed at the Department of Clinical Microbiology, Odense University Hospital from January 1st 2017 - December 31st 2020

Exclusion Criteria:

* Primary care physicians with a postal code in an area of Funen Island with a Lyme neuroborreliosis incidens of < 4.7/100.000

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of days from symptom debut to beginning of antibiotic treatment for Lyme neuroborreliosis | 0-90 days
  Number of days from debut of neurological symptoms to beginning of antibiotic treatment for Lyme neuroborreliosis.

SECONDARY OUTCOMES:
Number of yearly referred Lyme patients | Up to 4 years (1460 days).
  Number of yearly referred patients in the two study arms in the two years before the intervention (2017+2018) and after the intervention (2019+2020).
Number of Borrelia antibody tests in peripheral blood ordered by primary care physicians | Up to 4 years (1460 days).
  Number of Borrelia antibody tests in peripheral blood ordered by primary Health care physicians in the two study arms in the two years before (2017+2018) and after (2019 + 2020) the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrikke C Knudtzen, MD, Principal Investigator — Department of Infectious Diseases, Odense University Hospital
Locations (1):
- Clinical Center for Emerging and Vectorborne Infections, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to Denmark´s strict data-sharing Laws, data will not be shared after completion of study.

REFERENCES:
- [Result] Knudtzen FC, Andersen NS, Jensen TG, Skarphedinsson S. Characteristics and Clinical Outcome of Lyme Neuroborreliosis in a High Endemic Area, 1995-2014: A Retrospective Cohort Study in Denmark. Clin Infect Dis. 2017 Oct 16;65(9):1489-1495. doi: 10.1093/cid/cix568. PMID 29048514
- [Derived] Knudtzen FC, Jensen TG, Andersen NS, Johansen IS, Hovius JW, Skarphedinsson S. An intervention in general practice to improve the management of Lyme borreliosis in Denmark. Eur J Public Health. 2022 Jun 1;32(3):436-442. doi: 10.1093/eurpub/ckac013. PMID 35323885